CLINICAL TRIAL: NCT07120685
Title: Proof of Concept in the Prevention of Post-bariatric Sarcopenia: Simulated Activation of the "Gravitostat", Randomized Pilot Study
Brief Title: Proof of Concept in the Prevention of Post-bariatric Sarcopenia: Simulated Activation of the "Gravitostat"
Acronym: GRAVITOSARC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AOI 2023 BOIRIE
Record Dates: First submitted 2025-07-09; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: Obesity &Amp; Overweight; Bariatric Surgery
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gravitostatic group (with mechanical load involving the use of a weighted vest) (Experimental)
  Interventions: Other: maintaining mechanical load
- Non-gravitostatic group (control group) (No Intervention)

INTERVENTIONS:
Other: maintaining mechanical load — The method for maintaining mechanical load (artificially reproducing the stabilization of initial body weight) will involve the use of a weighted vest.
  Participants will be asked to wear the weighted vest for at least eight hours a day over a four-week period without changing their lifestyle. Patients will also be contacted by phone every week after surgery to confirm that they are using the vest in accordance with the protocol and to collect information on any potential adverse events. During these calls, weight adjustments-based on body weight changes-will be discussed with the patient and regularly recorded to stay as close as possible to the initial body weight, with a tolerance of ±1 kg. However, the maximum weight of the vest will not exceed 15% of the patient's initial weight (weight at the time of surgery).
  Between the 4th and 12th week, patients will be asked to wear the weighted vest loaded with the "weight lost" calculated at week 4 for at least four hours per day.
  Arms: Gravitostatic group (with mechanical load involving the use of a weighted vest)

SUMMARY:
Due to its mechanical and metabolic functions, muscle loss leads to resistance to weight loss during caloric restriction, particularly in patients with obesity. The recent discovery of a "gravitational" homeostatic system, induced by an additional load to body weight, suggests the existence of a new weight control mechanism. Such a "gravitostat" would ensure a form of weight homeostasis mediated by afferent signals originating from osteocytes in response to gravity perception. This hypothesis, initially derived from animal studies, has more recently been tested in humans. It shows that "activation of the gravitostat" through artificial increases in body weight facilitates body weight reduction without affecting lean mass (LM). Therefore, this "gravitostat" could contribute to preserving LM despite the loss of fat mass , whereas its decline may compromise muscle mass and function after bariatric surgery, despite undeniable improvements in comorbidities.

The present study aims to reduce the "metabolic load" (i.e., decreasing insulin resistance and inflammation) to promote muscle protein anabolism, while maintaining the "mechanical load" (by preserving initial body weight during weight loss induced by bariatric surgery) in order to activate the "gravitostat" and preserve muscle mass and function.

Currently, there are no clear recommendations or strategies to prevent muscle loss in patients who have undergone bariatric surgery. This simple concept, applied during drastic muscle loss, should help improve muscle health.

ELIGIBILITY:
Inclusion Criteria:

* Female participants
* Aged between 18 and 60 years
* Planned for bariatric surgery, such as sleeve gastrectomy
* Able to give informed consent to participate in research
* Affiliated to a social security scheme

Exclusion Criteria:

* Women weighing 170 kg or more
* Inability to move around independently.
* Participants with a spinal pathology.
* Pregnant or breast-feeding women.
* Inability to comply with protocol recommendations.
* Adults under legal guardianship (curatorship, guardianship, deprivation of liberty, patients benefiting from a judicial protection measure or safeguard of justice).
* Refusal to participate.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Loss of lean mass at 1 monts and 3 months after bariatric surgery in patients undergoing "weight compensation" compared to a group of patients following a conventional approach (without gravitostat activation). | 1 month and 3 months after bariatric surgery
  lean mass measurement with dual energy x-ray absorptiometry, DXA

SECONDARY OUTCOMES:
Loss of lean mass at 6 months after bariatric surgery in patients undergoing "weight compensation" compared to a group of patients following a conventional approach (without gravitostat activation). | 6 months after bariatric surgery
  lean mass measurement with dual energy x-ray absorptiometry, DXA
Change from baseline on weight at 1 month (M1), 3 months (M3), and 6 months (M6) | 1 month (M1), 3 months (M3), and 6 months (M6)
Change from baseline on BMI at 1 month (M1), 3 months (M3), and 6 months (M6) | 1 month (M1), 3 months (M3), and 6 months (M6)
Change from baseline on waist circumference at 1 month (M1), 3 months (M3), and 6 months (M6) | 1 month (M1), 3 months (M3), and 6 months (M6)
Change from baseline on hip circumference at 1 month (M1), 3 months (M3), and 6 months (M6) | 1 month (M1), 3 months (M3), and 6 months (M6)
Muscle mass in the arms and legs at 1 month (M1), 3 months (M3), and 6 months (M6) after surgery | 1 month (M1), 3 months (M3), and 6 months (M6)
Changes in muscle function (Handgrip strength test) at 1 month (M1), 3 months (M3), and 6 months (M6) after surgery | 1 month (M1), 3 months (M3), and 6 months (M6)
Changes in muscle function (Short Physical Performance Battery (SPPB)) at 1 month (M1), 3 months (M3), and 6 months (M6) after surgery | 1 month (M1), 3 months (M3), and 6 months (M6)
Changes in muscle function (6-minute walk test (TM6)) at 1 month (M1), 3 months (M3), and 6 months (M6) after surgery | 1 month (M1), 3 months (M3), and 6 months (M6)
Changes from baseline on muscle architechture at 1 month (M1), 3 months (M3), and 6 months (M6) after surgery | 1 month (M1), 3 months (M3), and 6 months (M6)
  Analysis of muscle architecture and lipid infiltration using muscle ultrasound
Changes from baseline on bone architechture at 1 month (M1), 3 months (M3), and 6 months (M6) after surgery | 1 month (M1), 3 months (M3), and 6 months (M6)
  Analysis of bone mineral density (BMD) of trabecular and cortical bone compartments using peripheral quantitative computed tomography (PQCT)
Changes from baseline on bone architecture at 1 month (M1), 3 months (M3), and 6 months (M6) after surgery | 1 month (M1), 3 months (M3), and 6 months (M6)
  Analysis of bone strength of trabecular and cortical bone compartments using peripheral quantitative computed tomography (PQCT)
Changes from baseline on bone architecture at 1 month (M1), 3 months (M3), and 6 months (M6) after surgery | 1 month (M1), 3 months (M3), and 6 months (M6)
  Analysis of geometric parameters (volume, air) of trabecular and cortical bone compartments using peripheral quantitative computed tomography (PQCT)
Change from baseline on blood glucose at 1 month (M1), 3 months (M3), and 6 months (M6) after surgery | 1 month (M1), 3 months (M3), and 6 months (M6)
Change from baseline on cholesterol at 1 month (M1), 3 months (M3), and 6 months (M6) after surgery | 1 month (M1), 3 months (M3), and 6 months (M6)
Change from baseline on triglycerides at 1 month (M1), 3 months (M3), and 6 months (M6) after surgery | 1 month (M1), 3 months (M3), and 6 months (M6)
Change from baseline on insulin levels at 1 month (M1), 3 months (M3), and 6 months (M6) after surgery | 1 month (M1), 3 months (M3), and 6 months (M6)
Change from baseline on CRP at 1 month (M1), 3 months (M3), and 6 months (M6) after surgery | 1 month (M1), 3 months (M3), and 6 months (M6)
Change from baseline on urinary creatinine at 1 month (M1), 3 months (M3), and 6 months (M6) after surgery | 1 month (M1), 3 months (M3), and 6 months (M6)
Effect of weight compensation at 1 month (M1), 3 months (M3), and 6 months (M6) after surgery on Plasma, serum, and urinary biomarkers | 1 month (M1), 3 months (M3), and 6 months (M6)
  Biological collection
Effect on Maximal strength | 1 month (M1), 3 months (M3), and 6 months (M6)
  Effect of weight compensation at 1 month (M1), 3 months (M3), and 6 months (M6) after surgery on maximum strenght (isokinetic dynamometry)
Effect on Food intake | 1 month (M1), 3 months (M3), and 6 months (M6)
  Effect of weight compensation at 1 month (M1), 3 months (M3), and 6 months (M6) after surgery on Food intake (nutrient intake using the "Nutrilog" software)
Effect of weight compensation at 1 month (M1), 3 months (M3), and 6 months (M6) after surgery on Nitrogen balance | 1 month (M1), 3 months (M3), and 6 months (M6)
Effect on Quality of life using a visual analog scale | 1 month (M1), 3 months (M3), and 6 months (M6)
  Effect of weight compensation at 1 month (M1), 3 months (M3), and 6 months (M6) after surgery on Quality of life using a visual analog scale
Effect on Food preferences and reward | 1 month (M1), 3 months (M3), and 6 months (M6)
  Effect of weight compensation at 1 month (M1), 3 months (M3), and 6 months (M6) after surgery on Food preferences and reward by using LFPQ (Leeds Food Preference Questionnaire)
To assess the effect of weight compensation at 1 month (M1), 3 months (M3), and 6 months (M6) after surgery on energy expenditure | 1 month (M1), 3 months (M3), and 6 months (M6)
  Energy expenditure (resting and total)
Effect on substrate utilization during an incremental submaximal walking exercise at 1 month (M1), 3 months (M3), and 6 months (M6) after surgery on energy expenditure | 1 month (M1), 3 months (M3), and 6 months (M6)
  Evaluate the use of energy substrates through the oxidation of carbohydrates and lipids an incremental submaximal walking exercise using in indirect calorimetry.
Effect on perceived exertion during an exercise (Borg scale) | 1 month (M1), 3 months (M3), and 6 months (M6)
  Effect of weight compensation at 1 month (M1), 3 months (M3), and 6 months (M6) after surgery on perceived exertion during an incremental submaximal walking exercise
Effect of heart rate | 1 month (M1), 3 months (M3), and 6 months (M6)
  During an incremental submaximal walking exercise
Effect of weight compensation on spontaneous physical activity using accelerometry | on day 4 or the day after returning home following surgery, and then at 1 month (M1) and 3 months (M3) after surgery.
  Effect of weight compensation on spontaneous physical activity (sedentary, low, moderate and intense) per day (min/d) at baseline, on day 4 or the day after returning home following surgery, and then at 1 month (M1) and 3 months (M3) after surgery.
Study the longitudinal evolution of weight every week until M1, then every 2 weeks until M3 for the experimental group. | every week until 1st month, then every 2 weeks until 3rd month after bariatric surgery
Study the longitudinal evolution of BMI every week until M1, then every 2 weeks until M3 for the experimental group. | every week until 1st month, then every 2 weeks until 3rd month after bariatric surgery
Tolerance with wearing the vest for the experimental group | from bariatric surgery to the end at 3 months
  Tolerance with wearing the vest for the experimental group, using a patient diary.
Compliance with wearing the vest for the experimental group | from bariatric surgery to the end at 3 months
  Compliance with wearing the vest for the experimental group, using a patient diary.

CONTACTS AND LOCATIONS:
Overall Officials: Yves BOIRIE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ciangura C, Bouillot JL, Lloret-Linares C, Poitou C, Veyrie N, Basdevant A, Oppert JM. Dynamics of change in total and regional body composition after gastric bypass in obese patients. Obesity (Silver Spring). 2010 Apr;18(4):760-5. doi: 10.1038/oby.2009.348. Epub 2009 Oct 15. PMID 19834464
- [Background] Thivel D, Boirie Y. The Gravitostat theory: Body fat is lost but is fat-free mass preserved? EClinicalMedicine. 2020 Oct 3;27:100531. doi: 10.1016/j.eclinm.2020.100531. eCollection 2020 Oct. No abstract available. PMID 33033796
- [Background] Ohlsson C, Hagg DA, Hammarhjelm F, Dalmau Gasull A, Bellman J, Windahl SH, Palsdottir V, Jansson JO. The Gravitostat Regulates Fat Mass in Obese Male Mice While Leptin Regulates Fat Mass in Lean Male Mice. Endocrinology. 2018 Jul 1;159(7):2676-2682. doi: 10.1210/en.2018-00307. PMID 29800288
- [Background] Jansson JO, Palsdottir V, Hagg DA, Schele E, Dickson SL, Anesten F, Bake T, Montelius M, Bellman J, Johansson ME, Cone RD, Drucker DJ, Wu J, Aleksic B, Tornqvist AE, Sjogren K, Gustafsson JA, Windahl SH, Ohlsson C. Body weight homeostat that regulates fat mass independently of leptin in rats and mice. Proc Natl Acad Sci U S A. 2018 Jan 9;115(2):427-432. doi: 10.1073/pnas.1715687114. Epub 2017 Dec 26. PMID 29279372